CLINICAL TRIAL: NCT04296500
Title: Herbal Medicine for Inflammatory Bowel Diseases: a Development of Pattern Identification Algorithm by Retrospective Analysis of Case Series Data
Brief Title: A Development of Inflammatory Bowel Disease Pattern Identification Algorithm Using Case Series Data
Status: Completed | Type: Observational
Sponsor: Hyangsook Lee, KMD, PhD (Other)
Responsible Party: Sponsor-Investigator, Hyangsook Lee, KMD, PhD, Professor, Kyunghee University
Organization: Kyunghee University (Other)
Other Study IDs: KyungheeU
Record Dates: First submitted 2020-03-03; First posted 2020-03-05 (Actual); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: Inflammatory Bowel Diseases
Keywords: Herbal prescription; Herbal medicine; Pattern identification; Algorithm; Decision tree; TF-IDF
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Decision tree algorithm training/testing: The investigators divided data of 67 patients into 5 groups to do 5 fold cross validation. Four groups were used to train decision tree algorithm and one group was used to test it.
  Interventions: Other: Decision tree modeling

INTERVENTIONS:
Other: Decision tree modeling — A decision tree analysis was employed to explore the process of decision-making on types of pattern based on the existence or nonexistence of a symptom. At the end of tree presented is the proportion of patients who are categorised into each pattern.
  In this study, the classification was performed by applying the classification and regression tree (CART) algorithm using Scikit-learn package of Python, which performs a division using the Gini coefficient or the decrement of dispersion. The Gini coefficient is one of the tools for measuring entropy or diversity in each node and it measures the decrement by comparing the information entropy before and after separation. To avoid overfitting, the maximum number of leaf nodes was limited to four and the pruning method which complied with the principle of minimum description length was applied.

SUMMARY:
This study aimed to identify inflammatory bowel disease (IBD) patterns based on presenting symptoms and to suggest algorithms for determining pattern and herbal prescriptions for corresponding patterns. The investigators collected symptom data of 67 IBD patients who achieved and maintained clinical remissions after they had taken herbal medicine prescriptions. Prescriptions were categorised into 5 patterns, which were named after main features and symptoms of included patients. Associations between presenting symptoms and patterns were visualised using a term frequency inverse document frequency (TF-IDF) method. Determining IBD patterns from symptoms of patients was analysed and charted by decision tree modeling.

DETAILED DESCRIPTION:
Herbal prescriptions are one of the most sought complementary and alternative medicine treatment strategies for inflammatory bowel disease patients. However, variability in pattern identification of Traditional Chinese Medicine (TCM)/Traditional East Asian Medicine (TEAM) has been criticised. Using data of patients who achieved and maintained clinical remission after TCM/TEAM herbal medicine prescription, the investigators aimed to develop treatment algorithms refined by identified pattern and key symptoms which practitioners can easily discriminate.

Based on herbal prescriptions which induced clinical remission, IBD patients were divided into 5 patterns, i.e., Large intestine type, Water-dampness type, Respiratory type, Upper gastrointestinal (GI) tract type, and Coldness type. By term frequency-inverse document frequency (TF-IDF) method, the association between 22 symptoms that were described as indications of the herbal medicine prescriptions and 5 patterns were analysed. Decision tree modeling was used for prediction of relevant patterns from symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of IBD by gastroenterologist
* Patients have achieved and maintained clinical remission of IBD symptoms after they took herbal prescriptions
* Patients have provided written informed consent

Exclusion Criteria:

* Details regarding any of 25 symptoms were omitted

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who had been diagnosed with IBD by gastroenterologist and achieved clinical remission after treatment with herbal medicine prescriptions
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2007-11-01 (Actual); Primary Completion 2015-02-28 (Actual); Study Completion 2015-10-28 (Actual)

PRIMARY OUTCOMES:
Accuracy of pattern identification algorithm | Oct 2015
  Pattern identification algorithm was suggested using a decision tree method. Decision tree method was employed to explore the process of decision making on types of pattern based on clinical features of patients.

CONTACTS AND LOCATIONS:
Overall Officials: Hyangsook Lee, Doctor, Principal Investigator — Kyunghee University
Locations (1):
- Acupuncture & Meridian Science Research Centre, Seoul, South Korea

REFERENCES:
- [Background] Bernstein CN, Fried M, Krabshuis JH, Cohen H, Eliakim R, Fedail S, Gearry R, Goh KL, Hamid S, Khan AG, LeMair AW, Malfertheiner, Ouyang Q, Rey JF, Sood A, Steinwurz F, Thomsen OO, Thomson A, Watermeyer G. World Gastroenterology Organization Practice Guidelines for the diagnosis and management of IBD in 2010. Inflamm Bowel Dis. 2010 Jan;16(1):112-24. doi: 10.1002/ibd.21048. PMID 19653289
- [Background] Panaccione R, Rutgeerts P, Sandborn WJ, Feagan B, Schreiber S, Ghosh S. Review article: treatment algorithms to maximize remission and minimize corticosteroid dependence in patients with inflammatory bowel disease. Aliment Pharmacol Ther. 2008 Sep 15;28(6):674-88. doi: 10.1111/j.1365-2036.2008.03753.x. PMID 18532990
- [Background] Abitbol V, Lahmek P, Buisson A, Olympie A, Poupardin C, Chaussade S, Lesgourgues B, Nahon S. Impact of complementary and alternative medicine on the quality of life in inflammatory bowel disease: results from a French national survey. Eur J Gastroenterol Hepatol. 2014 Mar;26(3):288-94. doi: 10.1097/MEG.0000000000000040. PMID 24407360
- [Background] Lee MS, Lee JA, Alraek T, Bian ZX, Birch S, Goto H, Jung J, Kao ST, Moon SK, Park B, Park KM, You S, Yun KJ, Zaslawski C. Current research and future directions in pattern identification: Results of an international symposium. Chin J Integr Med. 2016 Dec;22(12):947-955. doi: 10.1007/s11655-014-1833-3. Epub 2014 Jun 18. PMID 24938445
- [Background] Yu F, Takahashi T, Moriya J, Kawaura K, Yamakawa J, Kusaka K, Itoh T, Morimoto S, Yamaguchi N, Kanda T. Traditional Chinese medicine and Kampo: a review from the distant past for the future. J Int Med Res. 2006 May-Jun;34(3):231-9. doi: 10.1177/147323000603400301. PMID 16866016
- [Background] Liu B, Zhou X, Wang Y, Hu J, He L, Zhang R, Chen S, Guo Y. Data processing and analysis in real-world traditional Chinese medicine clinical data: challenges and approaches. Stat Med. 2012 Mar 30;31(7):653-60. doi: 10.1002/sim.4417. Epub 2011 Dec 9. PMID 22161304